CLINICAL TRIAL: NCT00901459
Title: A Controlled Laboratory Study of the Effects on Cue-Induced Craving in Dependent Smokers
Acronym: rTMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00002339
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2012-12

CONDITIONS: Nicotine Dependence
Keywords: Repetitive Transcranial Magnetic Stimulation; Cigarette Smoker; Cigarette Dependence; To block cue-elicited craving in dependent cigarette smokers
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rTMS 90% MT - Low frequency rTMS (Active Comparator): Intervention type: device. Intervention description: low frequency rTMS was administered over the superior frontal gyrus (SFG) during the presentation of smoking and control cues using 90% MT (Motor Threshold) 1 Hz rTMS Dose on Superior Frontal Gyrus
  Interventions: Device: Active rTMS Condition
- Location Control (Active Comparator): rTMS Dosing: 90% MT (Motor Threshold) 1 Hz rTNS Location: Motor Cortex
  Interventions: Device: rTMS Location Control Condition
- Frequency Control (Active Comparator): rTMS Dosing: 90% MT (Motor Threshold) 10 Hz rTNS Location: Superior Frontal Gyrus
  Interventions: Device: rTMS Frequency Control Condition

INTERVENTIONS:
Device: Active rTMS Condition — Low frequency rTMS (90% Motor Threshold at 1 HZ) will be administered over the superior frontal gyrus (SFG) during the presentation of smoking and control cues.
  Arms: rTMS 90% MT - Low frequency rTMS
Device: rTMS Location Control Condition — Low frequency rTMS (90% Motor Threshold at 1 HZ) will be administered over the motor cortex (MC) during the presentation of smoking and control cues.
  Arms: Location Control
Device: rTMS Frequency Control Condition — High frequency rTMS (90% Motor Threshold at 10 HZ) will be administered over the superior frontal gyrus (SFG) during the presentation of smoking and control cues.
  Arms: Frequency Control

SUMMARY:
The purpose of this study is to investigate the use of repetitive transcranial magnetic stimulation (rTMS) to block craving for cigarettes in smokers. rTMS is an investigational procedure, where a device called a "stimulator" provides electricity to a device that creates a magnetic field. This device is placed against the scalp in the front of the head so that the magnetic field is focused on an area of the brain that is thought to be involved in craving for cigarettes. rTMS is an investigational procedure so therefore being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA). Changes in magnetic fields during rTMS administration change electrical currents which may affect brain activity and function.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the effects of rTMS on cue-induced craving in dependent smokers. We hypothesize that low frequency rTMS over the SFG will block cue-induced craving. In order to test this hypothesis, subjects will undergo three conditions:

1. active condition: low frequency rTMS was administered over the superior frontal gyrus (SFG) during the presentation of smoking and control cues
2. location control condition: low frequency rTMS was administered over motor cortex (MC) during the presentation of smoking and control cues
3. frequency control condition: high frequency rTMS was administered over the SFG during the presentation of smoking and control cues

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 50 years of age;
2. dependent smoker of > 10 cigarettes per day of cigarettes yielding >0.5mg nicotine (by Federal Trade Commission rated yields);
3. have smoked cigarettes for at least three cumulative years;
4. an afternoon carbon monoxide reading of at least 10ppm;
5. be in general good health based on physical examination, EKG, serum chemistries, CBC, and urinalysis and
6. show evidence of greater craving following exposure to in vivo smoking versus control cues

Exclusion Criteria:

1. Individuals with a clinically defined neurological disorder or insult including, but not limited to, any condition likely to be associated with increased intracranial pressure;
2. space occupying brain lesion;
3. any history of seizure EXCEPT those therapeutically induced by ECT (Electro Convulsive Therapy);
4. history of cerebrovascular accident;
5. transient ischemic attack within two years;
6. cerebral aneurysm;
7. dementia;
8. Parkinson's disease;
9. Huntington's chorea;
10. multiple sclerosis;
11. current lung disease or lung disorder;
12. hypertension (systolic >140 mmHg, diastolic > 90 mmHg);
13. hypotension (< 90 mmHg, diastolic < 60 mmHg);
14. coronary artery disease;
15. cardiac rhythm disorder;
16. impaired hepatic or renal function (based on documented diagnosis or abnormal chemistries) except gallstones or kidney stones;
17. other major medical or psychiatric condition;
18. use of any concurrent hypertensive, psychiatric, or psychoactive medication;
19. any concurrent medication that lowers seizure threshold;
20. smokeless tobacco, pipe, or cigar use in the past 30 days;
21. nicotine replacement therapy, or other smoking cessation therapy within the past 30 days;
22. increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head trauma with loss of consciousness for > 5 minutes;
23. ECT treatment within 3 months prior to screening visit;
24. failure to respond to ECT treatment (i.e., consistent with ATHF level 2 or higher);
25. a true positive response to any question on the Transcranial Magnetic Stimulation Adult Safety Screen questionnaire;
26. history of treatment with rTMS therapy for any disorder;
27. use of any investigational drug within 30 days of the screening visit;
28. history of treatment with Vagus Nerve Stimulation;
29. use of any medication(s) with active CNS properties within 1 week of the screening visit;
30. cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease; intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
31. known or suspected pregnancy;
32. positive urine drug screen or reported drug abuse in the past 30 days;
33. clinically significant laboratory abnormality, in the opinion of the investigator or study physician;
34. women who are breast-feeding; women of child-bearing potential not using a medically accepted form of contraception when engaging in sexual intercourse;
35. current chronic pain or other pain condition that interferes with daily activities or requires use of prescription medication;
36. claustrophobia or abnormal fear of cramped or confined space;
37. Individuals where a motor threshold response is not elicited with stimulation at or below 80% of maximum output;
38. active ulcer within the past 30 days;
39. frequent migraines (great than four in the past 30 days);
40. Females who score greater than or equal to 13 and males who score greater than or equal to 15 on the AUDIT (Alcohol Use Disorders Identification Test)will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University; Andrew D Krystal, M.D., M.S., Principal Investigator — Duke University; Francis J McClernon, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Center for Nicotine & Smoking Cessation Research, Durham, North Carolina, United States

REFERENCES:
- [Derived] Rose JE, McClernon FJ, Froeliger B, Behm FM, Preud'homme X, Krystal AD. Repetitive transcranial magnetic stimulation of the superior frontal gyrus modulates craving for cigarettes. Biol Psychiatry. 2011 Oct 15;70(8):794-799. doi: 10.1016/j.biopsych.2011.05.031. Epub 2011 Jul 18. PMID 21762878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was consented on 5/12/2009 and the final participant on 6/22/2010 at the Duke Center for Nicotine and Smoking Cessation Research. During the recruitment phase of the study 148 potential subjects were consented and 7 read the consent form and chose not to participate.
Pre-assignment Details: Of the 148 participants that were consented for this study only 21 subjects met study criteria the others were excluded from participation for the following reasons:
  70-Did Not Meet Inclusion Criteria 6-Lab Results 6-Lost to Contact 26-Medical 14-Met exclusion criteria 3-Refused to participate 2-Unable To Meet Study Requirements
Groups:
- All Study Participants: Active:
  rTMS Dosing: 90% MT (Motor Threshold) 1 Hz rTMS Location: Superior Frontal Gyrus
  Location Control:
  rTMS Dosing: 90% MT (Motor Threshold) 1 Hz rTMS Location: Motor Cortex
  Frequency Control:
  rTMS Dosing: 90% MT (Motor Threshold) 10 Hz rTNS Location: Superior Frontal Gyrus
Period: Overall Study
Arm/Group | All Study Participants
Started | 21
Completed | 15
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.9 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Craving for Cigarettes After Smoking Cues Versus Neutral Cues Using a Repeated Measure Design.
Description: Cigarette craving was assessed orally during each rTMS Session, before and after each stimulus presentation and cigarette smoking with a brief version of the Shiffman-Jarvik questionnaire (14), which contained items assessing cigarette craving using the following subscale: CRAVING ("urges to smoke," "miss a cigarette," and "crave cigarettes"), MOOD ("calm," "tense," and "irritable"), AROUSAL ("wide awake," "able to concentrate"), and HUNGER ("feel hungry"). The scale for the Shiffman-Jarvik questionnaire is a Likert item scale with measurements 1-Not at All; 2-Very Little; 3-A Little; 4-Moderately; 5- A Lot; 6-Quite A Lot and 7-Extremely. The change in craving for cigarettes after smoking cues versus neutral cues using the parenthetical items listed above with the subscale CRAVING were used to determine the primary outcome. A negative value represents a decrease in reported cigarette craving.
Time Frame: Following exposure to in vivo cues
Population: A repeated measures design exposed participants to three different rTMS conditions over 3 separate visits, with order counterbalanced using latin square design.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Active: rTMS Dosing: 90% MT (Motor Threshold) 1 Hz rTMS Location: Superior Frontal Gyrus
- Location Control: rTMS Dosing: 90% MT (Motor Threshold) 1 Hz rTMS Location: Motor Cortex
- Frequency Control: rTMS Dosing: 90% MT (Motor Threshold) 10 Hz rTMS Location: Superior Frontal Gyrus
Arm/Group | Active | Location Control | Frequency Control
Number analyzed (Participants) | 15 | 15 | 15
units on a scale | -.18 (.95) | .12 (1.30) | 1.29 (1.52)
Statistical Analysis 1: Comparison: Active vs Frequency Control; A pairwise t-test was performed to contrast the active rTMS condition with the frequency control condition; Test type: Superiority or Other; p = 0.014, t-test, 2 sided — A Holm correction to p values was made to control for type 1 error; df=14; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [0.51 to 2.43], Standard Error of Mean 0.44 — The parameter estimated is the difference in craving change between smoking cues and neutral cues in the 10Hz sfg condition (Frequency control)and the corresponding craving change in the 1Hz sfg condition (active)
Statistical Analysis 2: Comparison: Active vs Location Control; A pairwise t-test was performed to contrast the active rTMS condition with the location control condition; Test type: Superiority or Other; p = 0.49, t-test, 2 sided; df=13; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.64 to 1.22], Standard Error of Mean 0.4 — The parameter estimated is the difference in craving change between smoking cues and neutral cues in the 1Hz sfg condition (active)and the corresponding craving change in the 1Hz moc condition (location control)
Statistical Analysis 3: Comparison: Location Control vs Frequency Control; A pairwise t-test was performed to contrast the location control rTMS condition with the frequency control condition; Test type: Superiority or Other; p = 0.09, t-test, 2 sided — A Holm correction to p values was made to control for type 1 error; df=13; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [0.52 to 1.39], Standard Error of Mean 0.44 — The parameter estimated is the difference in craving change between smoking cues and neutral cues in the 10Hz sfg condition (frequency control)and the corresponding craving change in the 1Hz moc condition (location control)

2. Secondary Outcome: Change in Craving for Cigarettes After Controlled Smoke Presentations.
Description: Craving reduction was assessed orally by an item on the cigarette evaluation questionnaire ("Did it immediately reduce your craving for cigarettes?") after smoking presentations through the controlled puff volume apparatus.
Time Frame: After smoking a cigarette through the controlled puff volume apparatus during rTMS
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active: rTMS Dosing: 90% MT (Motor Threshold) 1 Hz rTNS Location: Superior Frontal Gyrus
Arm/Group | Active | Location Control | Frequency Control
Number analyzed (Participants) | 15 | 14 | 15
units on a scale | -.18 (.95) | .12 (1.30) | 1.29 (1.52)

ADVERSE EVENTS:
Arm/Group | Active | Location Control | Frequency Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes